CLINICAL TRIAL: NCT01395680
Title: Trajectories of Regenerating Family Resilience in Adolescents With Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 201105004RC
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-06

CONDITIONS: Cancer
Keywords: cancer adolescent; resilience
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cancer adolescent

SUMMARY:
Family resilience is an important strength to help family to manage life challenge successfully, and to reorganize family function. However, few studies have showed the trajectory of family resilience in adolescents with cancer over time. The purposes of this study are to know the trend of family resilience in adolescents with cancer from previous 3 months to the first year of newly diagnosed, and to examine the relationships among family members' stress, family satisfaction, and family resilience in adolescents with cancer.

DETAILED DESCRIPTION:
The inclusion criteria of adolescents with cancer are: 1) 12-20 years of age, 2) newly diagnosed with cancer about 3 months, 3) willing and able to complete own report questionnaires. The study is designed as repeated measurement. Considering attrition rate may be more than 60%. Therefore, of necessity, the proposed sample size was set at 60 families.

Data will be collected by a structured questionnaire (a demographic questionnaire and 4 scales). The study consists of four times of data collection time point as follows: approximately 3 month (t1), 6 months (t2), 9 months (t3), and 12 months (t4) after the diagnosis of cancer in adolescents. Each participant may take 20-30 minutes to finish the structured questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of adolescents with cancer are: 1) 12-20 years of age, 2) newly diagnosed with cancer about 3 months, 3) willing and able to complete own report questionnaires.

Exclusion Criteria:

* terminal stage

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: cancer adolescent aged 12-20 years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Tsamm Lin, MD, Principal Investigator — National Taiwan University Hospital,Taipei,Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan